CLINICAL TRIAL: NCT02216929
Title: The Demographics, Mortality and Clinical Diagnosis of the Patients Who Were Evaluated, Intubated and Interned to ICU by the Anesthesiology in 2010-2011
Brief Title: Assessment of the Patients of Emergency Consultation
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Gulsah Karaoren (Other Government)
Responsible Party: Sponsor-Investigator, Gulsah Karaoren, Doctor, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Other Study IDs: GK2
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2011-01

CONDITIONS: Demographics of Intubated Patients Due to an Urgent Call
Keywords: intubation; intensive care; withholding treatment; cancer; terminal care; APACHE
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The demographic data, mortality rates and clinical diagnoses of the patients who were evaluated, intubated and interned to ICU by the anesthesiology department due to an urgent consultation call from the emergency department in 2010-2011.

Primary outcome: an examination of demographic data, predicted mortality rates and the clinical diagnosis of the patients Secondary outcome: to determine the terminal cancer ratio Inclusion criteria: patients throughout the hole hospital whom was intubated by the anaesthesiology team due to an emergency consultation call Exclusion criteria: patients who refused treatment

DETAILED DESCRIPTION:
The demographic data and findings completed in the Emergency Department were obtained from the patient cards and information related to existing diseases was obtained from the patient records for the cases included in the study.

Predicted mortality values were calculated for each patient with Apache II and SAPS II values using the worst or most critical physiological and laboratory parameters in the first 24 hours in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* patients throughout the hole hospital whom was intubated by the anaesthesiology team due to an urgent consultation call

Exclusion criteria:

* patients who refused treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study aimed to retrospectively evaluate patients throughout the whole hospital who were intubated and interned to the ICU by anaesthesiology team due to an urgent consultation call in our hospital during 2010-2011.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The evaluation of the terminal phase cancer ratio | 12 months
  To determine the ratio of patients with terminal phase cancer who were intubated and interned to the intensive care unit.

SECONDARY OUTCOMES:
Demographic data of urgent anaesthesiology consultations required intubation | 12 months
  The evaluation of the demographics, clinical diagnosis and the calculated values of APACHE II, SAPS II and predicted mortality of the patients who were intubated and interned to the ICU by anesthesiology department due to an urgent consultation call.

OTHER OUTCOMES:
The ratio of patients required cardiopulmonary resuscitation | 12 months
  The rate of CPR, the APACHE II and SAPS II expanded values of the patients required CPR .

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Oz, Prof Dr, Study Director — Medipol University Faculty of Medicine
Locations (1):
- Istanbul University Faculty of Cerrahpasa Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kim AS, Youn CH, Ko HJ, Kim HM. The survival time of terminal cancer patients: prediction based on clinical parameters and simple prognostic scores. J Palliat Care. 2014 Spring;30(1):24-31. PMID 24826440
- [Background] Uy J, White DB, Mohan D, Arnold RM, Barnato AE. Physicians' decision-making roles for an acutely unstable critically and terminally ill patient. Crit Care Med. 2013 Jun;41(6):1511-7. doi: 10.1097/CCM.0b013e318287f0dd. PMID 23552510
- [Result] Lissauer ME, Naranjo LS, Kirchoffner J, Scalea TM, Johnson SB. Patient characteristics associated with end-of-life decision making in critically ill surgical patients. J Am Coll Surg. 2011 Dec;213(6):766-70. doi: 10.1016/j.jamcollsurg.2011.09.003. PMID 22107920